CLINICAL TRIAL: NCT03436576
Title: Comparison of Autologous Serum 20% and Autologous Serum 50% for the Treatment of Severe Dry Eye
Brief Title: Efficacy of Two Concentrations of Autologous Serum for the Treatment of Severe Dry Eye
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Hospital Dr Sotero del Rio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SERUM2050
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Dry Eye; Keratoconjunctivitis Sicca; Sjogren's Syndrome; Corneal Diseases; Conjunctival Diseases; Keratitis; Lacrimal Apparatus Diseases
Keywords: Autologous serum; Concentration; Autologous serum 20%; Autologous serum 50%; Severe dry eye
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca; Sjogren's Syndrome; Corneal Diseases; Conjunctival Diseases; Keratitis; Lacrimal Apparatus Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous Serum 20% (Active Comparator): Treatment with Autologous Serum 20% for 2 months
  Interventions: Drug: Autologous Serum 20%
- Autologous Serum 50% (Active Comparator): Treatment with Autologous Serum 50% for 2 months
  Interventions: Drug: Autologous Serum 50%

INTERVENTIONS:
Drug: Autologous Serum 20% — Instillation of 1 drop of Autologous Serum 20% four times a day
  Other Names: Autologus serum low concentration
  Arms: Autologous Serum 20%
Drug: Autologous Serum 50% — Instillation of 1 drop of Autologous Serum 50% four times a day
  Other Names: Autologus serum high concentration
  Arms: Autologous Serum 50%

SUMMARY:
The purpose of this study is to compare the effects of autologous serum 20% and autologous serum 50% for the treatment of Severe Dry Eye Syndrome

DETAILED DESCRIPTION:
To determine the difference between autologous serum 20% vs 50%, in terms of improvement of symptoms, improvement of ocular surface parameters and acceptable tolerability in patients with severe dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Man/woman ≥ 18 years old, able to freely give consent to participate in the study
* At least 1 of the following tests altered:

  * Ocular Surface Disease Index (OSDI) Test symptoms > 32
  * BUT ≤5 seconds
  * Oxford staining ≥ 3
  * Schirmer Test without anesthesia ≤ 5 mm

Exclusion Criteria:

* Sensitivity or known intolerance to any of the products used in the study
* Contraindication of venipuncture
* Story of ocular infections within the 6 previous months to study inclusion
* Any active ocular pathology other than Dry Eye Syndrome
* Use of contact lenses in the 3 previous months to study inclusion
* No pregnant or breastfeeding women is allowed to participate in the study. Childbearing potential women must use contraceptive means during the whole study.
* Participation in another clinical trial in the last 30 days before study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-12 (Estimated); Primary Completion 2018-10-19 (Estimated); Study Completion 2018-11-19 (Estimated)

PRIMARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI) Score | 1 month
  The Ocular Surface Disease Index (OSDI) is a 12-item questionnaire designed to provide a rapid assessment of the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning.
  The overall OSDI score defines the ocular surface as normal (0-12 points) or as having mild (13-22 points), moderate (23-32 points), or severe (33-100 points) disease.

SECONDARY OUTCOMES:
Change in Tear Break Up Time (TBUT) | 1 week, 1 month, 2 months
  The TBUT is based on the time of tear rupture after the instillation of fluorescein.
  The shorter the time of rupture, the greater the tear dysfunction
Change in Oxford Staining score | 1 week, 1 month, 2 months
  The Oxford scale is based on the amount of ocular surface (cornea and conjunctiva) that is stained with lysine or green fluorescein. The severity of the staining points is classified into 6 stages (0-5) from absent to marked epithelial damage.
Change in Schirmer I | 1 week, 1 month, 2 months
  It is a tear production test. The Schirmer I test is performed without anesthesia. Two thin strips of filter paper (Whatman 5mm x 35mm) are placed on the bottom of the lower conjunctival sac at the junction of the middle third and the outer third to prevent injury to the cornea. It is recommended to ask the subject to keep their eyes closed to limit the effect of blinking. The strips are kept positioned for 5 minutes and then they are removed and the amount that was moistened is read, in mm.
  The lower the value, the greater the deficit of tear production
Change in Ocular Surface Disease Index (OSDI) Score | 1 week, 2 months
  The Ocular Surface Disease Index (OSDI) is a 12-item questionnaire designed to provide a rapid assessment of the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning.
  The overall OSDI score defines the ocular surface as normal (0-12 points) or as having mild (13-22 points), moderate (23-32 points), or severe (33-100 points) disease.

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Liberman, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Dr. Sótero del Río, Puente Alto, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No